CLINICAL TRIAL: NCT07195331
Title: Reduced Dose vs Standard Dose of Indocyanine Green in Near-infrared Fluorescence Cholangiography During Laparoscopic Cholecystectomy: a Randomized Clinical Trial.
Brief Title: Comparison Between Standard and Reduced Doses of Indocyanine Green in Fluorescence Cholangiography During Laparoscopic Cholecystectomy.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low-DOTIG; 2025-522535-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-04; First posted 2025-09-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Cholecystectomy Surgery
Keywords: laparoscopic cholecystectomy; bile ducts; cholangiography; indocyanine green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.5 mg >3h before surgery (Experimental)
  Interventions: Drug: Intravenous injection of indocianine green at least three hours before surgery at a dose of 2.5 mg per subject.
- 0.25 mg 15-30 min before surgery (Experimental)
  Interventions: Drug: Intravenous injection of indocianine green 15 to 30 minutes before surgery at a dose of 0.25 mg per subject.

INTERVENTIONS:
Drug: Intravenous injection of indocianine green at least three hours before surgery at a dose of 2.5 mg per subject. — A dilution will be prepared by dissolving 25 mg of ICG in 10 mL of water for injectable solutions, yielding a concentration of 2.5 mg/mL. Once the solution is prepared, 1 mL will be administered directly via a peripheral venous line in the patient's upper limb.
  Arms: 2.5 mg >3h before surgery
Drug: Intravenous injection of indocianine green 15 to 30 minutes before surgery at a dose of 0.25 mg per subject. — A dilution will be prepared by dissolving 25 mg of ICG in 25 mL of water for injectable solutions, yielding a concentration of 1 mg/mL. Subsequently, 0.25 mL will be administered as a direct intravenous injection via a peripheral venous line in the patient's upper limb.
  Arms: 0.25 mg 15-30 min before surgery

SUMMARY:
Introduction:

This protocol outlines a randomized phase IV clinical trial designed to compare the efficacy of two different doses of indocyanine green (ICG) used in near-infrared fluorescent cholangiography during laparoscopic cholecystectomy (LC)-the current gold standard treatment for symptomatic cholelithiasis. Despite its effectiveness, LC is still associated with significant risks, particularly bile duct injury (BDI), a severe complication that this study aims to mitigate.

Phase: Phase IV Study design: Multicenter, randomized, open-label, parallel-group clinical trial (modified intention-to-treat).

Objectives:

Primary objective:

* To analyze differences between treatment groups (standard dose 2.5 mg >3h preoperative vs reduced dose 0.25 mg immediate preoperative 15-30 min) during laparoscopic cholecystectomy in:
* Visualization of extrahepatic biliary structures
* Degree of visualization
* Degree of background liver fluorescence interference
* Perceived utility of the technique

Secondary objectives:

* Influence of BMI, biliary pathology type, surgery type, prior inflammation, surgical difficulty, previous instrumentation, and laparoscopic imaging system on results
* Intraoperative and postoperative complication rates
* 30-day mortality
* Impact on operative time and hospital stay
* Correlation between subjective and objective fluorescence assessment (ducts-to-liver fluorescence ratio) Population: Patients ≥18 years indicated for laparoscopic cholecystectomy (elective, early or urgent deferred).

Main inclusion criteria:

* Age ≥18 years
* Signed informed consent
* Indication for laparoscopic cholecystectomy (symptomatic cholelithiasis, gallbladder polyps with surgical indication)

Main exclusion criteria:

* Age <18 years
* Pregnancy or lactation
* Chronic kidney disease (stage >IIIb)
* ICG or iodinated contrast allergy
* Functional thyroid disease
* Emergency non-deferrable surgery
* Open approach
* Suspicion of gallbladder carcinoma
* Inability to understand the study Investigational product: Indocyanine green (ICG), intravenous administration

This multicenter study involves two hospitals in Castilla y León, Spain, and plans to enroll 122 adult patients meeting specific clinical criteria for LC. Participants will be randomized into two treatment arms and will receive ICG accordingly:

* Group 1: 2.5 mg >3h before surgery
* Group 2: 0.25 mg 15-30 min before surgery Fluorescence will be assessed both subjectively by the surgical team and objectively through digital image analysis using specialized software to calculate the bile duct-to-liver fluorescence ratio (RFBH).

Endpoints:

* Rates and degree of biliary structure identification pre- and post-dissection
* Perceived utility of cholangiography
* Liver background fluorescence interference
* Ducts-to-liver fluorescence ratio Duration: 12 months recruitment + 1 month follow-up = total 13 months Countries: Spain Ethics: The study will be conducted in accordance with ICH-GCP, EU Clinical Trials Regulation No 536/2014, and applicable national regulations.

Beyond comparing the diagnostic performance of two dosing strategies, this study seeks to provide evidence supporting a more practical and logistically feasible approach for implementing ICG fluorescence cholangiography in routine surgical practice, without compromising diagnostic accuracy or patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Signed informed consent.
* Indication for laparoscopic cholecystectomy (symptomatic cholelithiasis or gallbladder polyps).

Exclusion Criteria:

* Age <18 years.
* Pregnancy or lactation.
* Chronic kidney disease (stage >IIIb).
* ICG allergy.
* Allergy to other iodinated contrast
* Functional thyroid disease.
* Emergency non-deferrable surgery.
* Open approach.
* Suspicion of gallbladder cancer.
* Inability to understand the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification of biliary structures prior to dissection of the hepatocystic triangle. | During surgery
  The identification of extrahepatic biliary structures prior to the dissection of the hepatocystic triangle is defined as the visualization of fluorescence emitted by these structures during laparoscopic surgery, at a minimum distance of 15 cm from the anatomical structure and with a perpendicular orientation of the laparoscopic optics to it. The following scale will be used: Category 1. Identification of the cystic duct prior to dissection Category 2. Identification of the common bile duct prior to dissection Category 3. Identification of the junction of the cystic duct with the common bile duct prior to dissection Category 4. Identification of the union of the cystic duct with the gallbladder prior to dissection Category 5. Identification of the common hepatic duct prior to dissection Category 6. Identification of biliary anatomical variables prior to dissection.
Identification rate of biliary structures after dissection of the hepatocystic triangle | During surgery.
  The identification of extrahepatic biliary structures after dissection of the hepatocystic triangle is defined as the visualization of fluorescence emitted by these structures during laparoscopic surgery, at a minimum distance of 15 cm from the anatomical structure and with a perpendicular orientation of the laparoscopic optics over it. The following scale will be used: Category 1. Identification of the cystic duct after the dissection Category 2. Identification of the common bile duct after the dissection. Category 3. Identification of the junction of the cystic duct with the common bile duct after the dissection Category 4. Identification of the union of the cystic duct with the gallbladder after the dissection Category 5. Identification of the common hepatic duct after the dissection Category 6. Identification of biliary anatomical variables after the dissection.
Degree of identification of extrahepatic biliary structures prior to dissection of the hepatocystic triangle | During surgery
  The degree of identification of extrahepatic biliary structures is assessed using a 3-point Likert scale:
  Poor (1): unable to distinguish fluorescence in extrahepatic biliary structures.
  Good (2): able to visualize fluorescence at least in the main bile duct. Excellent (3): able to visualize fluorescence in the main bile duct, the cystic duct, and their junction.
  The assessment of this variable must be performed before any surgical maneuver within the hepatocystic triangle.
Degree of identification of extrahepatic biliary structures after dissection of the hepatocystic triangle | During surgery.
  The degree of identification of extrahepatic biliary structures is assessed using a 3-point Likert scale:
  Poor (1): unable to distinguish fluorescence in extrahepatic biliary structures.
  Good (2): able to visualize fluorescence at least in the main bile duct. Excellent (3): able to visualize fluorescence in the main bile duct, the cystic duct, and their junction.
  The assessment of this variable must be performed before any surgical maneuver within the hepatocystic triangle.
Perceived usefulness of fluorescence cholangiography (FC). | During surgery
  The usefulness of FC during surgery is assessed using a 3-point Likert scale:
  Not useful (1): the technique did not provide any benefit or even hindered the procedure.
  Moderately useful (2): the technique guided certain phases of the procedure. Very useful (3): the technique guided most phases of the procedure, assisted decision-making, or even modified a previous surgical decision.
Degree to which background liver fluorescence (contrast between the liver and biliary ducts) was perceived as disturbing | During surgery
  The disturbing effect of background liver fluorescence is assessed using a 3-point Likert scale:
  None (0): liver fluorescence was almost imperceptible and/or allowed clear visualization of hepatocystic triangle structures before dissection.
  Slightly disturbing (1): liver fluorescence was evident but still allowed clear visualization of hepatocystic triangle structures after dissection.
  Very disturbing (2): liver fluorescence was significantly disturbing and prevented identification of extrahepatic biliary anatomy either before or after dissection of the hepatocystic triangle.

SECONDARY OUTCOMES:
To analyze the rate of postoperative complications related to FC during LC. | From surgery to 30 days post-surgery
  The evaluation will be focused on identifying and quantifying adverse events potentially attributable to the use of fluorescence cholangiography (FC) during laparoscopic cholecystectomy (LC). Complications of interest will include, but will not be limited to, allergic reactions to indocyanine green, bile duct injury, postoperative bile leak, surgical site infection, or any other event directly associated with the intraoperative use of FC. The rate of these complications will be recorded and analyzed to assess the safety profile of FC as an adjunct to LC.
To analyze hospital and 30-day mortality rates. | From surgery to 30 days post-surgery
  Hospital and 30-day mortality rates will be assessed as key safety outcomes. Mortality is defined as any death occurring during the index hospital admission or within 30 days after laparoscopic cholecystectomy, regardless of cause. Both in-hospital and 30-day mortality will be systematically recorded to provide a comprehensive evaluation of short-term survival and to ensure patient safety in the context of fluorescence cholangiography use.
To analyze the impact of the technique on operative time, intraoperative/postoperative complications, and hospital stay. | From surgery to 30 days post-surgery.
  The impact of the technique on operative time, intraoperative and postoperative complications, and length of hospital stay will be analyzed. Operative time will be measured from the initial skin incision to wound closure. Intraoperative and postoperative complications will be prospectively recorded and categorized according to standardized surgical criteria. Length of hospital stay will be calculated in days from surgery until discharge. This analysis will allow evaluation of the overall clinical impact of the technique on surgical efficiency, patient outcomes, and resource utilization.
To analyze the correlation between the subjective and objective assessment of the procedure through the use of the bile duct-to-liver fluorescence ratio. | During surgery.
  In this trial, in addition to the subjective assessment of fluorescence, an objective evaluation will be introduced as a novel approach, with the aim of establishing a correlation between the two. For this purpose, the biliary duct-to-liver fluorescence ratio (BDHR) will be calculated by determining the average intensity in the biliary ducts and the average intensity in the hepatic tissue given by the fluorescense detected in the images taken during the procedure: BDHR=Intensity biliary duct/Intensity liver.
  The results will be interpreted as follows:
  BDHR = 1: Biliary duct fluorescence similar to hepatic parenchyma.
  BDHR > 1: Biliary duct fluorescence greater than hepatic parenchyma → Adequate visualization.
  BDHR < 1: Biliary duct fluorescence lower than hepatic parenchyma → Inadequate visualization.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime López, Medical Degree in Surgery, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA); Eva Alonso, Principal Investigator — Complejo Asistencial de Zamora.
Locations (2):
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Virgen de la Concha, Zamora, Zamora

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF